CLINICAL TRIAL: NCT01855867
Title: A Phase IV Open-label Evaluation of Safety, Tolerability and Acceptability of Elvitegravir / Cobicistat / Emtricitabine / Tenofovir Disoproxil Fumarate Single-tablet Regimen for Non-occupational Prophylaxis Following Potential Exposure to HIV-1
Brief Title: HIV Non-Occupational Post-Exposure Prophylaxis
Acronym: QUAD
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kenneth H. Mayer, MD (Other)
Collaborators: Gilead Sciences (Industry)
Responsible Party: Sponsor-Investigator, Kenneth H. Mayer, MD, Medical Director, The Fenway Institute, Fenway Community Health
Organization: Fenway Community Health (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: QUAD; IND: 116,967 (Other: FDA)
Record Dates: First submitted 2013-05-02; First posted 2013-05-17 (Estimated); Results first posted 2022-04-19 (Actual); Last update posted 2022-04-19 (Actual); Status verified 2022-03

CONDITIONS: Human Immunodeficiency Virus
Keywords: HIV; PEP; nPEP; Prophylaxis; Post Exposure Prophylaxis; exposure to HIV; HIV prevention
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Emtricitabine; Tenofovir; Elvitegravir, Cobicistat, Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Stribild (Other): Single dose Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg) taken for 28 days, within 72 hours of a possible sexual exposure to HIV
  Interventions: Drug: Single Dose Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg)

INTERVENTIONS:
Drug: Single Dose Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg)
  Other Names: Stribild; QUAD

SUMMARY:
The purpose of this study is to see if an anti-HIV medication known as Stribild (elvitegravir/cobicistat/emtricitabine/tenofovir DF) is safe, tolerable and acceptable when taken for 28 days, once a day after a possible, sexual, exposure to the Human Immune Deficiency Virus (HIV).

DETAILED DESCRIPTION:
Stribild is a combination of 1 integrase strand transfer inhibitor, 1 pharmacokinetic enhancer, and 2 nucleos(t)ide analog HIV-1 reverse transcriptase inhibitors, and was approved in August 2012, as a complete treatment regimen for HIV-1 infection in adults who are antiretroviral treatment-naïve. We are proposing to evaluate the safety, tolerability and acceptability of Stribild given to participants over age 18 after a possible sexual exposure to HIV-1. Enrolled participants will have experienced a moderate to high risk exposure, as outlined in the study protocol, within the last 72 hours - per 2005 Center for Disease Control and Prevention guidelines. Participants will take one Stribild tablet, by mouth, once a day for 28 days. Study staff will assess for changes in blood chemistries and clinical signs and symptoms from baseline health. Study participation is 90 days and will include HIV testing, STI screening, HIV/STI risk reduction counseling, clinical assessments, blood draws and surveys designed to gather knowledge and perception of HIV post-exposure prophylaxis (PEP) and HIV pre-exposure prophylaxis (PrEP). Conditional referrals to continued HIV/STI risk reduction counseling and testing will be made if risk remains high at study termination. In addition, participants will be connected to a medical provider if risk demonstrates a potential need for HIV pre-exposure prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* > Age of 18 at time of first visit.
* HIV uninfected on the basis of a negative HIV Rapid Test
* Willing and able to provide written informed consent.
* Willing and able to provide adequate locator information.
* Willing and able to return to all study visits.
* Willing to participate in all study procedures.
* Biologic women of childbearing potential: Willing to use contraception for as long as they are on study medication plus 7 days after.
* Possible sexual exposure to HIV-1, recent enough to permit receiving the first dose of study medication within 72 hours from the end of the exposure.

possible exposure could include:

1. Unprotected anal, vaginal, oral, or mucosal (e.g. conjunctival) exposure to ejaculate from a partner who is HIV-1 infected or high risk for HIV infection and of unknown HIV-1 serostatus (may include protected sexual exposure with condom failure, breakage or slippage); or
2. Unprotected penile exposure to cervicovaginal secretions or anorectal secretions from a partner who is HIV-1 infected or high risk for HIV infection and of unknown HIV-1 serostatus (may include protected sexual exposure with condom failure, breakage or slippage)

Exclusion Criteria:

* An active psychiatric illness or active drug or alcohol abuse that, in the opinion of the investigator, could prevent compliance with study procedures.
* Pregnancy and/or Breastfeeding.
* Biologic women who are actively trying to become pregnant.
* Acute or Chronic Hepatitis B infection, by history
* Acute or Chronic Renal Disease, by history
* Creatinine Clearance at or below 70mL/min (Cockcroft-Gault equation, Actual Weight)
* Known intolerance or allergy to tenofovir DF, emtricitabine, elvitegravir or cobicistat
* Currently taking or plans to take prohibited medication while enrolled in the study.

  * Prohibited Medications*

    * Propulsid (Cisapride)
    * UroXatral (Alfuzosin)
    * Dihydroergotamine
    * Ergotamine
    * Methylergonovine
    * St John's Wort (Hypericum perforatum)
    * Altocor, Altoprev, Mevacor (Lovastatin)
    * Zocor (Simvastatin)
    * Orap (Pimozide)
    * Rifadin, Rimactane (Rifampin)
    * Viagra (Sildenafil when dosed as REVATIO)
    * Halcion (Triazolam)
    * Versed (Midazolam) (when administered orally)
    * Antiretroviral medications used to treat or prevent HIV infection.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-05; Primary Completion 2014-04 (Actual); Study Completion 2016-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth H. Mayer, MD, Principal Investigator — The Fenway Institute, Fenway Community Health
Locations (1):
- Fenway Community Health, Boston, Massachusetts, United States

REFERENCES:
- See also: 2005 CDC Guidelines on Antiretroviral Postexposure Prophylaxis After Sexual, Injection-Drug Use, or Other Nonoccupational Exposure to HIV in the United States — http://www.cdc.gov/mmwr/preview/mmwrhtml/rr5402a1.htm

RESULTS

PARTICIPANT FLOW:
Groups:
- Stribild: Coformulated Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg) taken for 28 days, within 72 hours of a possible sexual exposure to HIV
  Coformulated Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg)
Period: Overall Study
Arm/Group | Stribild
Started | 100
Completed | 100
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Stribild
Number analyzed (Participants) | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 100
  >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 34.1 [19 to 62]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 98
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 12
  Not Hispanic or Latino | 88
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 8
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 9
  White | 83
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 100

OUTCOME MEASURES:

1. Primary Outcome: Number of Adverse Event Occurrences
Description: The number of adverse events reported
Time Frame: 90 days
Population: 100 participants were enrolled
Measure: Number; unit: events
Arm/Group | Stribild
Number analyzed (Participants) | 100
events
  Diarrhea | 38
  Fatigue | 28
  Nausea/Vomiting | 28
  Headache | 14
  Dizziness/Lightheadness | 6
  Body Aches/Muscle and Joint Pain | 2

2. Secondary Outcome: Number of Participants With Self-Reported Missed Doses
Description: self-reported missed doses
Time Frame: Day 30
Measure: Count of Participants; unit: Participants
Arm/Group | Stribild
Number analyzed (Participants) | 100
Participants | 29
Statistical Analysis 1: Comparison: Stribild; using historical controls; Test type: Superiority — Statistical significance was determined at the alpha 0.05 level. The study regimen completion rates of participants in the current study taking a fixed dose once daily combination of elvitegravir/cobicistat/TDF/FTC were compared to historical controls who used PEP regimens consisting of TDF/FTC daily and raltegravir twice daily, or earlier regimens of twice daily zidovudine (AZT)/lamivudine (3TC) and a protease inhibitor, using chi-square tests for independence; p < 0.05, Chi-squared — Reported p-value was calculated, and is not attempting to indicate the threshold for statistical significance; chi square

3. Other Pre Specified Outcome: nPEP Failure (HIV Infection During Study Participation)
Description: nPEP failure, meaning HIV infection during study participation, as measured during HIV testing at day 0, day 30 and day 90
Time Frame: 90 days
Measure: Number; unit: reactive test
Groups:
- Stribild: Coformulated Elivitegravir (150mg), Combicistat (150mg), Emtricitabine (200mg), Tenofovir DF (300mg) taken for 28 days, within 72 hours of a possible sexual exposure to HIV
Arm/Group | Stribild
Number analyzed (Participants) | 100
reactive test | 0

ADVERSE EVENTS:
Time Frame: 90 days
Arm/Group | Stribild
All-Cause Mortality (participants affected / at risk) | 0/100
Serious Adverse Events (participants affected / at risk) | 0/100
Other Adverse Events (participants affected / at risk) | 91/100
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stribild (N=100)
Diarrhea (Gastrointestinal disorders) | 38 (38)
Fatigue (Nervous system disorders) | 28 (28)
Nausea/vomiting (Gastrointestinal disorders) | 28 (28)
headache (Nervous system disorders) | 18 (18)
dizziness/lightheadedness (Nervous system disorders) | 6 (6)
body/muscle/joint aches (Musculoskeletal and connective tissue disorders) | 2 (2) — pain or overall discomfort

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No